CLINICAL TRIAL: NCT02742987
Title: CLOpidogrel Versus TIcagreLor for Antiplatelet Maintenance in DIAbetic Patients Treated With Percutaneous Coronary Intervention: Results of the CLOTILDIA Study
Brief Title: Clopidogrel Versus Ticagrelor in Type-2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Germano Di Sciascio, Prof. Germano Di Sciascio, Campus Bio-Medico University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLOTILDIA
Record Dates: First submitted 2016-03-24; First posted 2016-04-19 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-07

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor group (Experimental): Ticagrelor 90 mg twice daily + standard medical therapy
  Interventions: Drug: Ticagrelor; Drug: Standard medical therapy
- Clopidogrel group (Experimental): Clopidogrel 150 mg once daily + standard medical therapy
  Interventions: Drug: Clopidogrel; Drug: Standard medical therapy

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor 90 mg twice daily
  Arms: Ticagrelor group
Drug: Clopidogrel — Clopidogrel 150 mg once daily
  Arms: Clopidogrel group
Drug: Standard medical therapy — Standard medical therapy for patients with coronary artery disease undergoing percutaneous coronary interventions

SUMMARY:
CLOTILDIA is a single-center, prospective, randomized, open label, cross-over study evaluating the effects of ticagrelor versus high-dose clopidogrel on endothelial function and platelet reactivity in patients with type-2 diabetes mellitus (T2DM) treated with percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* stable coronary disease
* coronary revascularization with PCI at least 1 month prior to recruitment

Exclusion Criteria:

* acute coronary syndrome
* platelet count <70x109/l
* active bleeding or bleeding diathesis
* history of intracranial bleeding
* gastrointestinal bleeding <6 months
* cerebrovascular accident <3 months
* history of malignancy
* concomitant need for oral anticoagulant therapy
* severe liver disease or chronic renal failure (glomerular filtration rate <30 ml/min /1.73m2)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ticagrelor Group | Clopidogrel Group
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor Group | Clopidogrel Group | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (9.5) | 67.7 (8.1) | 66.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 19 | 18 | 37
Region of Enrollment [Number; unit: participants]
  Italy | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Flow-mediated Dilation of the Brachial Artery
Description: Percent dilation of the brachial artery, as assessed with vascular ultrasound, from baseline to post-occlusion
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: FMD (%)
Arm/Group | Ticagrelor Group | Clopidogrel Group
Number analyzed (Participants) | 21 | 21
FMD (%) | 16.6 (4.8) | 11.6 (3.9)

2. Secondary Outcome: Number of Patients With Flow-mediated Dilation of the Brachial Artery <7%
Time Frame: 4 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Endothelium-independent Dilation of the Brachial Artery
Description: Percent dilation of the brachial artery, as assessed with vascular ultrasound, from baseline to post-administration of 0.5 mg sublingual nitroglycerin
Time Frame: 4 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Platelet Reactivity
Description: Platelet reactivity assessed with the VerifyNow P2Y12 Assay
Time Frame: 4 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Number of Patients With Platelet Reactivity >256 P2Y12 Reaction Units
Time Frame: 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Ticagrelor Group | Clopidogrel Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 1/21 | 0/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor Group (N=21) | Clopidogrel Group (N=21)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No